CLINICAL TRIAL: NCT02964091
Title: Simplifying Hepatitis C Antiviral Therapy in Rwanda for Elsewhere in the Developing World
Acronym: SHARED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Partners in Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHARED 092415
Record Dates: First submitted 2016-11-03; First posted 2016-11-15 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C Virus; sofosbuvir/ledipasvir; Efficacy
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Harvoni (Other): sofosbuvir/ledipasvir once daily for 12 weeks
  Interventions: Drug: sofosbuvir/ledipasvir

INTERVENTIONS:
Drug: sofosbuvir/ledipasvir
  Other Names: Harvoni

SUMMARY:
The main purpose of the study is to evaluate the efficacy, safety and tolerability of a medication, ledipasvir/sofosbuvir (LDV/SOF), used to treat individuals with chronic hepatitis C virus (HCV) in Rwandan adults. A sub-cohort of participants will have limited laboratory monitoring to determine the minimum laboratory tests necessary.

DETAILED DESCRIPTION:
This is an open-label single arm study that will evaluate the antiviral efficacy, safety and tolerability of ledipasvir/sofosbuvir fixed dose combination administered for 12 weeks in HCV treatment-naive and treatment-experienced participants with chronic genotype 1 or 4 HCV infection. Approximately 240 participants will be enrolled and treated with sofosbuvir (SOF) 400 mg/LDV 90 mg fixed dose combination (FDC) one tablet once daily for 12 weeks in the SHARED 1 study. Sixty additional participants will be enrolled in the SHARED 2 sub-cohort with laboratory monitoring blinded to study clinicians.

ELIGIBILITY:
Inclusion Criteria:

* patients that are willing and able to provide written informed consent
* age ≥ 18 years
* HCV RNA ≥ 103 IU/mL
* HCV genotype 1 or 4
* screening ultrasound excluding hepatocellular carcinoma (HCC)
* acceptable laboratory values (hemoglobin ≥8.0 g/dL, platelet count ≥40,000/mm3; AST, ALT, and alkaline phosphatase ≤10 × ULN; creatinine clearance ≥30 mL/min)
* general good health
* ability to comply with study procedures
* HIV-infected patients must have completed at least 6 months of any approved HIV antiretroviral therapy (ART) per Rwanda National Guidelines 2013, have been taking for at least 2 weeks prior to screening ART compatible with SOF/LDV (efavirenz, rilpivirine, raltegravir, dolutegravir, emtricitabine, lamivudine, zidovudine, tenofovir), have screening HIV RNA < 200 copies/mL, and have screening CD4 T-cell count of ≥100 cells/µL

Exclusion Criteria:

* current or history of clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage)
* active tuberculosis
* other clinically-significant illness (except HCV and/or HIV) or any other major medical disorder
* active Hepatitis B infection
* difficulty with blood collection and/or poor venous access for the purposes of phlebotomy
* any IFN-containing regimen within 8 weeks prior to screening or any prior exposure to HCV-specific direct-acting antiviral agent (other than a NS3/4A protease inhibitor and SOF), current pregnancy or breastfeeding, and active drug or alcohol use or dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with sustained viral response as defined by an HCV RNA below the limit of quantification 12 weeks after discontinuation of study treatment | After study completion (24 weeks)
  To determine the hepatitis C virus (HCV) antiviral efficacy of sofosbuvir/ledipasvir (SOF/LDV) fixed-dose combination (FDC) as measured by the proportion of participants with sustained viral response 12 weeks after discontinuation of study treatment (SVR12) in Rwanda.
Proportion of participants with sustained viral response as defined by an HCV RNA below the limit of quantification 12 weeks after discontinuation of study treatment, with limited lab monitoring | After study completion (24 weeks)
  To determine the HCV antiviral efficacy of SOF/LDV FDC, as measured by the proportion of participants with sustained viral response 12 weeks after discontinuation of study treatment (SVR12), with limited lab monitoring in Rwanda.
Proportion of participants with a new grade 3 or 4 adverse event or premature study drug discontinuation due to an adverse event. | After study completion (24 weeks)
  To evaluate the safety and tolerability of SOF/LDV FDC in Rwanda

SECONDARY OUTCOMES:
A set of minimum required monitoring tests | After study completion (24 weeks)
  A set of minimum required monitoring tests
Distribution of HCV genotypes subtypes among participants | After study completion (24 weeks)
  Distribution of HCV genotypes subtypes among participants
SVR12, stratified by genotypic subtype | After study completion (24 weeks)
  SVR12, stratified by genotypic subtype
Basic demographic and clinical characteristics of patients referred for HCV treatment | After study completion (24 weeks)
  Basic demographic and clinical characteristics of patients referred for HCV treatment
Adherence to SOF/LDV measured by pill count | After 12 weeks medication therapy
  Adherence to SOF/LDV measured by pill count
Proportion of participants with virologic failure | After study completion (24 weeks)
  Proportion of participants with virologic failure
Proportion of participants with HCV RNA below the level of quantitation (BLQ) while on treatment | After study completion (24 weeks)
  Proportion of participants with HCV RNA below the level of quantitation (BLQ) while on treatment
Proportion of HIV co-infected participants that maintain HIV-1 RNA< 200 copies/mL while on HCV treatment | After 12 weeks of medication therapy
  Proportion of HIV co-infected participants that maintain HIV-1 RNA< 200 copies/mL while on HCV treatment
Proportion of participants reporting increased quality of life after SVR12 using the Medical Outcomes Study HIV Health Survey | After study completion (24 weeks)
  To determine the effect of SOF/LDV and SVR12 on quality of life in Rwanda

CONTACTS AND LOCATIONS:
Overall Officials: Neil Gupta, MD, Principal Investigator — Partners in Health; Jules Kabahizi, MD, Principal Investigator — Rwanda Military Hospital; Aimable Mbituyumuremyi, MD, Principal Investigator — Rwanda Biomedical Centre; Philip Grant, MD, Principal Investigator — Stanford University; Claude M Muvunyi, MD, Principal Investigator — University of Rwanda
Locations (1):
- Rwanda Military Hospital, Kanombe, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, study data, data dictionary, data collection instruments, and informed consent forms are available upon request from the corresponding author. De-identifiable individual participant data will be made available 9 months after the publication date and ending 36 months after the publication date. Forms and data can be accessed by written request to the corresponding author and the study sponsor, Partners In Health. The data will be made available following evaluation and approval of proposed use by the study sponsor and signed data access agreement with the study sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identifiable individual participant data will be made available 9 months after the publication date and ending 36 months after the publication date.
Access Criteria: Forms and data can be accessed by written request to the corresponding author and the study sponsor, Partners In Health.
  The data will be made available following evaluation and approval of proposed use by the study sponsor and signed data access agreement with the study sponsor.

REFERENCES:
- [Derived] Gupta N, Mbituyumuremyi A, Kabahizi J, Ntaganda F, Muvunyi CM, Shumbusho F, Musabeyezu E, Mukabatsinda C, Ntirenganya C, Van Nuil JI, Kateera F, Camus G, Damascene MJ, Nsanzimana S, Mukherjee J, Grant PM. Treatment of chronic hepatitis C virus infection in Rwanda with ledipasvir-sofosbuvir (SHARED): a single-arm trial. Lancet Gastroenterol Hepatol. 2019 Feb;4(2):119-126. doi: 10.1016/S2468-1253(18)30382-0. Epub 2018 Dec 11. PMID 30552056